CLINICAL TRIAL: NCT02008565
Title: Controlling Anal Incontinence by Performing Anal Exercises With Biofeedback or Loperamide (CAPABLe): a Randomized Placebo Controlled Trial
Brief Title: Controlling Anal Incontinence by Performing Anal Exercises With Biofeedback or Loperamide (CAPABLe)
Acronym: CAPABLe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: The Cleveland Clinic (Other); University of Alabama at Birmingham (Other); University of California, San Diego (Other); Duke University (Other); National Institutes of Health (NIH) (NIH); University of New Mexico (Other); Women and Infants Hospital of Rhode Island (Other); RTI International (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PFDN- 18PO1; 2U10HD041261 (NIH); 2U10HD054215 (NIH); 2U10HD041267 (NIH); 1U10HD069006 (NIH); 2U10HD054214 (NIH); 1U10HD069013 (NIH); 1U10HD069025 (NIH); 1U10HD069010 (NIH); 1U01HD069031 (NIH)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Loperamide; anal exercises; biofeedback
MeSH Terms: conditions — Fecal Incontinence | interventions — Loperamide; Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo - Exercise plus Biofeedback (Placebo Comparator): Placebo and biofeedback intervention. Placebo doses range from 2mg every other day to 8mg per day. Capsules are taken by mouth once a day for 24 weeks.
  Anal exercises with biofeedback intervention is a total of six sessions with trained personnel occurring every 2 weeks over a 12-week period. Sessions are held at the following study visits: baseline, 2, 4, 6, 9, and 12 week visits.
  Interventions: Drug: Placebo; Behavioral: Anal exercises with biofeedback
- Loperamide - Exercise plus Biofeedback (Experimental): Loperamide and biofeedback intervention. Loperamide doses range from 2mg every other day to 8mg per day. Capsules are taken by mouth once a day for 24 weeks.
  Anal exercises with biofeedback intervention is a total of six sessions with trained personnel occurring every 2 weeks over a 12-week period. Sessions are held at the following study visits: baseline, 2, 4, 6, 9, and 12 week visits.
  Interventions: Drug: Loperamide; Behavioral: Anal exercises with biofeedback
- Placebo - Education Only (Placebo Comparator): Placebo and education (usual care). Placebo doses range from 2mg every other day to 8mg per day. Capsules are taken by mouth once a day for 24 weeks.
  Participants receive education and a NIDDK Bowel Control Educational pamphlet.
  Interventions: Drug: Placebo; Behavioral: Usual Care
- Loperamide - Education Only (Experimental): Loperamide and education (usual care). Loperamide doses range from 2mg every other day to 8mg per day. Capsules are taken by mouth once a day for 24 weeks.
  Participants receive education and a NIDDK Bowel Control Educational pamphlet.
  Interventions: Drug: Loperamide; Behavioral: Usual Care

INTERVENTIONS:
Drug: Loperamide — Participants randomized to the loperamide group will begin with 2mg of loperamide/day. The participant will be administered the Patient Global Symptom Control rating scale (PGSC) to determine dose escalation. Participants who report inadequate control of stool leakage on the PGSC will be instructed to increase the daily dose of loperamide by 2 mg up to a maximum of 8 mg per day (1-4 capsules). Bothersome adverse events and resulting dose reduction will be based exclusively on the result of the Patient Global Tolerability Scale (PGTS). The daily dose will be decreased by 2mg to a minimum of 2mg every other day. If a PGSC score indicates inadequate control of stool leakage combined with a PGTS score indicating bothersome side effects, the participant will discontinue the study medication.
  Other Names: Imodium
  Arms: Loperamide - Education Only; Loperamide - Exercise plus Biofeedback
Drug: Placebo — Participants randomized to the placebo arm will begin the a dose of one capsule per day and will be dose increased or dose decreased using the same algorithm described for the loperamide arm.
  Other Names: Inactive Drug
  Arms: Placebo - Education Only; Placebo - Exercise plus Biofeedback
Behavioral: Anal exercises with biofeedback — Participants will receive a formal anal exercises training program that can be easily applied in an office setting with minimal participant burden. Participants will attend six anal exercises with biofeedback sessions with trained personnel over a 12-week period for the 24-week study. Sessions will include introduction, standard patient education, and exercises using anal manometry-assisted biofeedback introducing concepts such as shaping, generalization and termination. The protocol uses strength and sensory training including urge resistance training. During the final twelve weeks, participants will perform anal exercises on their own. The sessions with interventionists will occur every other week for 12 weeks (total 6 supervised sessions).
  Arms: Loperamide - Exercise plus Biofeedback; Placebo - Exercise plus Biofeedback
Behavioral: Usual Care — Usual care consists of patients receiving an educational pamphlet on fecal incontinence created by the National Institute of Diabetes and Digestive and Kidney Diseases.
  Arms: Loperamide - Education Only; Placebo - Education Only

SUMMARY:
The study is a multi-center, randomized, placebo controlled trial with participants randomized into one of four groups:

1. placebo/usual care (educational pamphlet)
2. loperamide/usual care (educational pamphlet)
3. placebo/anal exercises with biofeedback
4. loperamide/anal exercises with biofeedback

The primary outcome, change from baseline in St. Marks (Vaizey) Score at 24 weeks, will be compared between treatment groups using linear regression.

DETAILED DESCRIPTION:
The goals of this trial are to compare the use of loperamide to oral placebo and to compare the use of anal sphincter exercise training with biofeedback to usual care (educational pamphlet) in the treatment of women suffering from fecal incontinence (FI). We will test the following null hypotheses:

1. there is no difference in outcomes between women randomized to loperamide and women randomized to oral placebo for treatment of FI;
2. there is no difference in outcomes between women randomized to anal sphincter exercises with biofeedback and women randomized to usual care (educational pamphlet) for FI treatment;
3. there is no difference between women randomized to both treatments together and women randomized to either FI treatment alone; and
4. there is no correlation between anal manometry measurements and digital anal squeeze strength or measures of FI severity and bother.

A supplemental study, Stool Metabolome and Microbiome in Women with Fecal Incontinence in CAPABLe, will evaluate the stool metabolome and microbiome in women with fecal incontinence and unaffected age matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Fecal incontinence defined as any uncontrolled loss of liquid or solid fecal material that occurs at least monthly over the last 3 months that is bothersome enough to desire treatment

Exclusion Criteria:

* Stool consistency over the last 3 months that includes items 1 or 7 based on the Bristol Stool form scale
* Current or past diagnosis of colorectal or anal malignancy
* Diagnosis of inflammatory bowel disease
* Current or history of rectovaginal fistula or cloacal defect
* Rectal prolapse (mucosal or full thickness)
* Prior removal or diversion of any portion of colon or rectum
* Prior pelvic floor or abdominal radiation
* Refusal or inability to provide written consent
* Inability to conduct telephone interviews conducted in English or Spanish
* Fecal impaction by exam
* Untreated pelvic organ prolapse beyond the hymen; Patients with prolapse beyond the hymen who are currently using a pessary are eligible
* Incontinence only to flatus
* Has taken any loperamide (Imodium®) or diphenoxylate plus atropine (Lomotil®) in the last 30 days
* Previously received and failed treatment of fecal incontinence using loperamide (Imodium®) or diphenoxylate plus atropine (Lomotil®) over the last 3 months
* Current supervised anal sphincter exercise/pelvic floor muscle training with biofeedback
* Previously received and failed treatment of fecal incontinence using supervised anal sphincter exercise/pelvic floor muscle training with biofeedback
* Previous allergy or intolerance to loperamide
* Pregnant, nursing, or planning to become pregnant before the end of the study follow-up period.
* Childbirth within the last 3 months
* Currently taking anti-retroviral drugs
* Neurological disorders known to affect continence, including spinal cord injury, advanced multiple sclerosis or Parkinson's disease and debilitating stroke
* Known diagnosis of hepatic impairment
* Chronic abdominal pain in the absence of diarrhea

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J E Jelovsek, Study Chair — The Cleveland Clinic; Matthew Barber, Study Chair — The Cleveland Clinic
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, La Jolla, California
  - Kaiser San Diego, San Diego, California
  - University of New Mexico, Albuquerque, New Mexico
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown/Women and Infants Hospital of Rhode Island, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jelovsek JE, Markland AD, Whitehead WE, Barber MD, Newman DK, Rogers RG, Dyer K, Visco AG, Sutkin G, Zyczynski HM, Carper B, Meikle SF, Sung VW, Gantz MG; National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Controlling faecal incontinence in women by performing anal exercises with biofeedback or loperamide: a randomised clinical trial. Lancet Gastroenterol Hepatol. 2019 Sep;4(9):698-710. doi: 10.1016/S2468-1253(19)30193-1. Epub 2019 Jul 15. PMID 31320277

RESULTS

PARTICIPANT FLOW:
Groups:
- Loperamide - Exercise Plus Biofeedback: Participants receive loperamide drug and anal exercise with biofeedback intervention.
- Placebo - Exercise Plus Biofeedback: Participants receive placebo drug and anal exercise with biofeedback intervention.
- Loperamide - Education Only: Participants receive loperamide drug and educational pamphlet (usual care).
- Placebo - Education Only: Participants receive placebo drug and educational pamphlet (usual care).
Period: Overall Study
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Started | 86 | 84 | 88 | 42
Completed | 85 | 83 | 86 | 42
Not Completed | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Loperamide - Exercise Plus Biofeedback: Participants receive loperamide drug and anal exercises with biofeedback intervention.
- Placebo - Exercise Plus Biofeedback: Participants receive placebo drug and anal exercises with biofeedback intervention.
- Total: Total of all reporting groups
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only | Total
Number analyzed (Participants) | 85 | 83 | 86 | 42 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.9) | 63.2 (12.2) | 63.4 (10.6) | 62.6 (10.6) | 63.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 83 | 86 | 42 | 296
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 7 | 3 | 26
  Not Hispanic or Latino | 76 | 73 | 78 | 38 | 265
  Unknown or Not Reported | 1 | 2 | 1 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1 | 0 | 0 | 2 | 3
  Black/African American | 13 | 13 | 13 | 7 | 46
  More than one race | 4 | 1 | 0 | 0 | 5
  Other | 2 | 2 | 2 | 2 | 8
  White | 65 | 67 | 71 | 31 | 234
Vaginal deliveries, median [min, max] [Median (Full Range); unit: Vaginal deliveries] | 2.0 [0.0 to 7.0] | 2.0 [0.0 to 6.0] | 2.0 [0.0 to 6.0] | 2.0 [0.0 to 7.0] | 2.0 [0.0 to 7.0]
Cesarean deliveries, median [min, max] [Median (Full Range); unit: Cesarean deliveries] | 0.0 [0.0 to 4.0] | 0.0 [0.0 to 5.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 5.0]
Menstrual status, No. (%) [Count of Participants; unit: Participants]
  Not Sure | 2 | 7 | 5 | 2 | 16
  Post-menopausal | 74 | 69 | 74 | 34 | 251
  Pre-menopausal | 9 | 7 | 7 | 6 | 29
Currently using estrogen therapy, No. (%) [Count of Participants; unit: Participants]
  Oral/Patch | 7 | 8 | 10 | 3 | 28
  Vaginal | 24 | 22 | 19 | 10 | 75
  Not currently using estrogen therapy | 54 | 53 | 57 | 29 | 193
Current smoker, No. (%) [Count of Participants; unit: Participants]
  Current smoker | 3 | 8 | 8 | 2 | 21
  Not current smoker | 82 | 75 | 78 | 40 | 275
Connective tissue disease, No. (%) [Count of Participants; unit: Participants]
  Connective tissue disease | 3 | 5 | 3 | 1 | 12
  Does not have connective tissue disease | 82 | 78 | 83 | 41 | 284
Prior accidental bowel leakage surgery, No. (%) [Count of Participants; unit: Participants]
  Prior accidental bowel leakage surgery | 3 | 6 | 4 | 0 | 13
  No prior accidental bowel leakage surgery | 82 | 77 | 82 | 42 | 283
Prior rectal or anal surgery, No. (%) [Count of Participants; unit: Participants]
  Prior rectal or anal surgery | 13 | 11 | 9 | 7 | 40
  No prior rectal or anal surgery | 72 | 72 | 77 | 35 | 256
Prior hysterectomy, No. (%) [Count of Participants; unit: Participants]
  Prior hysterectomy | 45 | 40 | 45 | 18 | 148
  No prior hysterectomy | 40 | 43 | 41 | 24 | 148
Prior urinary incontinence surgery, No. (%) [Count of Participants; unit: Participants]
  Prior urinary incontinence surgery | 24 | 22 | 20 | 11 | 77
  No prior urinary incontinence surgery | 61 | 61 | 66 | 31 | 219
Prior pelvic organ prolapse surgery, No. (%) [Count of Participants; unit: Participants]
  Prior pelvic organ prolapse surgery | 22 | 22 | 18 | 8 | 70
  No prior pelvic organ prolapse surgery | 63 | 61 | 68 | 34 | 226
BMI, mean (SD) [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (7.4) | 28.5 (6.7) | 30.9 (6.6) | 30.5 (10.4) | 30.0 (7.8)
Bristol Stool Index, No. (%) [Count of Participants; unit: Participants]
  Type 2 (Sausage shaped but lumpy) | 18 | 9 | 7 | 11 | 45
  Type 3 (Like a sausage or snake but with cracks on | 12 | 11 | 17 | 3 | 43
  Type 4 (Like a sausage or snake, smooth and soft) | 21 | 28 | 29 | 15 | 93
  Type 5 (Soft blobs with clear cut edges) | 17 | 17 | 14 | 5 | 53
  Type 6 (Fluffy pieces with ragged edges, a mushy s | 17 | 18 | 19 | 8 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline St. Mark's (Vaizey) Score
Description: The primary outcome measure for all study arms is the change from baseline in St. Mark's (Vaizey) Score 24 weeks after treatment initiation to compare the marginal outcomes of anal exercise with biofeedback to usual care and loperamide to placebo.
  The St. Mark's (Vaizey) score, published in 1999, is commonly used in clinical studies and reports and was based on the Jorge-Wexner score but added two further items for assessment: the use of constipating medication and the presence of fecal urgency. Minimum score is 0 = perfect continence; maximum score is 24 = totally incontinent.
Time Frame: 12 and 24 weeks
Population: An intent-to-treat (ITT) analysis was performed for primary analyses. ITT analysis included all eligible participants who were randomized. The primary analyses included randomized patients who provided outcome data at 12 or 24 weeks.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 85 | 83 | 86 | 42
units on a scale
  12 Week St. Mark's Score: number analyzed (Participants) | 72 | 73 | 77 | 38
  12 Week St. Mark's Score | -5.5 [-7.2 to -3.9] | -4.4 [-6.0 to -2.8] | -4.5 [-6.1 to -2.9] | -3.4 [-6.0 to -0.8]
  24 Week St. Mark's Score: number analyzed (Participants) | 75 | 74 | 80 | 37
  24 Week St. Mark's Score | -9.7 [-11.9 to -7.5] | -5.9 [-8.1 to -3.7] | -6.2 [-8.1 to -4.2] | -4.5 [-7.1 to -1.9]
Statistical Analysis 1: Comparison: Loperamide - Exercise Plus Biofeedback vs Placebo - Exercise Plus Biofeedback; Test type: Superiority; p = 0.092, Mixed Models Analysis — significance assessed at type 1 error alpha=0.05; The models were adjusted for baseline Irritable Bowel Syndrome (IBS) status and clinical site

2. Secondary Outcome: Change in Quality of Life on Colorectal-Anal Distress Inventory (CRADI)
Description: The Pelvic Floor Distress Inventory is a 20-question, validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of an overall scale (range: 0-300) comprised of 3 sub-scales: 1) Pelvic Organ Prolapse Distress Inventory (range: 0-100), 2) Colorectal Anal Distress Inventory (range: 0-100), and 3) Urinary Distress Inventory (range: 0-100). The range of responses on the CRADI is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Scores are calculated by multiplying the mean value of all questions answered by 25 for the scale. The range of responses is: 0-100 with 0 (least distress) to 100 (most distress). Change = (Week [12, 24] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 85 | 83 | 86 | 42
units on a scale
  12 Week CRADI Score: number analyzed (Participants) | 71 | 72 | 72 | 37
  12 Week CRADI Score | -16.3 [-22.4 to -10.1] | -13.1 [-19.2 to -7.1] | -16.9 [-22.8 to -11.1] | -4.6 [-14.2 to 5.1]
  24 Week CRADI Score: number analyzed (Participants) | 72 | 70 | 74 | 35
  24 Week CRADI Score | -21.5 [-27.6 to -15.4] | -15.7 [-21.7 to -9.6] | -21.7 [-27.6 to -15.9] | -15.7 [-25.4 to -5.9]

3. Secondary Outcome: Change in Colorectal-Anal Subscale of the Pelvic Floor Impact Questionnaire Short Form (CRAIQ) Score
Description: The Pelvic Floor Impact Questionnaire short form (PFIQ-7) measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of 3 scales of 7 questions each: the Urinary Impact Questionnaire (UIQ; range 0-100), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; range 0-100), and the Colorectal-Anal Impact Questionnaire (CRAIQ; range 0-100). The range of responses on the CRAIQ is 0-3 with (0) Not at all, (1) Somewhat, (2) Moderately, and (3), Quite a bit. Scores are calculated by multiplying the mean value of all answered questions for a scale by 100 divided by 3. The range of responses is: 0-100 with 0 (least negative impact) to 100 (most negative impact). Change = (Week [12, 24] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 85 | 83 | 86 | 42
units on a scale
  12 Weeks: number analyzed (Participants) | 71 | 71 | 71 | 36
  12 Weeks | -12.5 [-18.5 to -6.4] | -10.8 [-16.8 to -4.9] | -15.8 [-21.6 to -9.9] | -12.3 [-21.9 to -2.8]
  24 Weeks: number analyzed (Participants) | 72 | 69 | 71 | 35
  24 Weeks | -41.3 [-57.9 to -24.6] | -32.4 [-48.8 to -15.9] | -41.6 [-57.8 to -25.4] | -17.3 [-26.9 to -7.8]

4. Secondary Outcome: Change From Baseline Accident-free Days at 12 and 24 Weeks
Description: Based on data collected from participant-completed diaries at baseline and 12 and 24 weeks, the outcome variable is computed as the difference in number of accident-free days at 12 and 24 weeks and the number of accident-free days at baseline. Only valid diaries were included in the analyses (e.g. completion of all 7 days for baseline and at least 3 complete days, not necessarily consecutive, for follow-up diaries).
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: accident-free days
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 85 | 82 | 85 | 41
accident-free days
  12 Weeks | 1.8 [1.1 to 2.5] | 1.9 [1.2 to 2.6] | 1.7 [1.0 to 2.4] | 1.4 [0.2 to 2.5]
  24 Weeks | 2.5 [1.8 to 3.2] | 1.9 [1.2 to 2.5] | 1.7 [1.0 to 2.4] | 2.1 [0.9 to 3.3]

5. Secondary Outcome: Change From Baseline Pad-change Leaks Per Day at 12 and 24 Weeks
Description: Based on data collected from participant-completed diaries at baseline and 12 and 24 weeks, the outcome variable is computed as the difference in number of fecal incontinence episodes per day resulting in a change in pad, clothes or underwear at 12 and 24 weeks and the number of fecal incontinence episodes resulting in a change in pad, clothes or underwear at baseline. Only valid diaries were included in the analyses (e.g. completion of all 7 days for baseline and at least 3 complete days, not necessarily consecutive, for follow-up diaries).
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pad-change leaks per day
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 85 | 82 | 85 | 41
pad-change leaks per day
  12 Weeks: number analyzed (Participants) | 73 | 73 | 71 | 37
  12 Weeks | -0.4 [-0.7 to -0.1] | -0.2 [-0.4 to 0.1] | -0.3 [-0.5 to 0.0] | -0.2 [-0.7 to 0.2]
  24 Weeks: number analyzed (Participants) | 71 | 72 | 78 | 35
  24 Weeks | -0.5 [-0.8 to -0.2] | -0.1 [-0.4 to 0.2] | -0.4 [-0.7 to -0.1] | -0.4 [-0.8 to 0.1]

6. Secondary Outcome: Change From Baseline Pad-change Leaks Per Week at 12 and 24 Weeks
Description: Based on data collected from participant-completed diaries at baseline and 12 and 24 weeks, the outcome variable is computed as the difference in number of fecal incontinence episodes per week resulting in a change in pad, clothes or underwear at 12 and 24 weeks and the number of fecal incontinence episodes resulting in a change in pad, clothes or underwear at baseline. Only valid diaries were included in the analyses (e.g. completion of all 7 days for baseline and at least 3 complete days, not necessarily consecutive, for follow-up diaries).
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pad-change leaks per week
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 85 | 82 | 85 | 41
pad-change leaks per week
  12 Weeks: number analyzed (Participants) | 73 | 73 | 71 | 37
  12 Weeks | -2.7 [-4.5 to -0.9] | -1.1 [-2.9 to 0.6] | -1.3 [-3.1 to 0.4] | -1.7 [-4.8 to 1.3]
  24 Weeks: number analyzed (Participants) | 71 | 72 | 78 | 35
  24 Weeks | -3.3 [-5.2 to -1.5] | -0.7 [-2.5 to 1.0] | -2.2 [-3.9 to -0.4] | -2.5 [-5.6 to 0.5]

7. Secondary Outcome: Change From Baseline Total Number of Leaks Per Day at 12 and 24 Weeks
Description: Based on data collected from participant-completed diaries at baseline and 12 and 24 weeks, the outcome variable is computed as the difference in daily average FI episodes at 12 and 24 weeks and the daily average FI episodes at baseline. Only valid diaries were included in the analyses (e.g. completion of all 7 days for baseline and at 3 complete days, not necessarily consecutive, for follow-up diaries).
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: leaks per day
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 85 | 82 | 85 | 41
leaks per day
  12 Weeks: number analyzed (Participants) | 73 | 73 | 71 | 37
  12 Weeks | -1.1 [-1.6 to -0.6] | -0.7 [-1.2 to -0.2] | -0.9 [-1.4 to -0.4] | -1.0 [-1.8 to -0.2]
  24 Weeks: number analyzed (Participants) | 71 | 72 | 78 | 35
  24 Weeks | -1.3 [-1.8 to -0.8] | -0.7 [-1.1 to -0.2] | -1.0 [-1.5 to -0.6] | -1.3 [-2.2 to -0.5]

8. Secondary Outcome: Change in Fecal Incontinence Severity Index (FISI) Score
Description: The Modified Manchester Health Questionnaire (MMHQ) includes the 4-item Fecal Incontinence Severity Index (FISI), which measures the severity of liquid, solid, mucus, or gas incontinence that occurs from "2 or more times per day," "once per day," "2 or more times per week," "once a week," to "1-3 times per month." Patient-weighted scores were used to determine severity and scores ranged from 0-61, with higher scores indicating worse fecal incontinence (FI) severity. An FISI score of 0 indicated continence.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 83 | 83 | 86 | 42
units on a scale
  12 Week MMHQ Severity Measures Score: number analyzed (Participants) | 69 | 70 | 66 | 34
  12 Week MMHQ Severity Measures Score | -12.4 [-19.0 to -5.8] | -10.6 [-17.1 to -4.0] | -14.4 [-20.8 to -7.9] | -7.8 [-18.5 to 2.8]
  24 Week MMHQ Severity Measures Score: number analyzed (Participants) | 70 | 67 | 66 | 34
  24 Week MMHQ Severity Measures Score | -19.1 [-25.7 to -12.5] | -15.0 [-21.6 to -8.4] | -19.2 [-25.7 to -12.7] | -20.0 [-30.5 to -9.5]

9. Secondary Outcome: Participants With Improvement in Patient Global Impression of Improvement (PGI-I) Score
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had improvement as indicated by a rating of 1 (very much better), 2 (much better), or 3 (a little better).
Time Frame: 12 and 24 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 83 | 81 | 84 | 41
Participants
  12 Weeks: number analyzed (Participants) | 71 | 72 | 72 | 37
  12 Weeks | 68 | 57 | 61 | 26
  24 Weeks: number analyzed (Participants) | 72 | 70 | 74 | 35
  24 Weeks | 67 | 59 | 60 | 25

10. Secondary Outcome: Change From Baseline Resting Anal Canal Pressures (mm of Hg) at 2 cm, 1 cm, and 0 cm Insertion at 12 and 24 Weeks
Description: Based on data collected from the manometry form, the outcome variable is computed as the difference in resting anal canal pressures (mm Hg) at 2 cm, 1 cm, and 0 cm insertion at 12 and 24 weeks and resting anal canal pressures (mm Hg) at 2 cm, 1 cm, and 0 cm insertion at baseline
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: resting anal canal pressure (mm Hg)
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 83 | 83 | 84 | 41
resting anal canal pressure (mm Hg)
  12 Week Maximum Anal Canal Pressure (Rest): number analyzed (Participants) | 68 | 69 | 76 | 37
  12 Week Maximum Anal Canal Pressure (Rest) | 52.6 [47.6 to 57.7] | 49.4 [44.4 to 54.4] | 51.1 [46.4 to 55.9] | 46.3 [38.5 to 54.2]
  24 Week Maximum Anal Canal Pressure (Rest): number analyzed (Participants) | 71 | 69 | 74 | 35
  24 Week Maximum Anal Canal Pressure (Rest) | 47.7 [42.7 to 52.7] | 47.8 [42.7 to 52.9] | 45.7 [40.8 to 50.5] | 46.5 [38.8 to 54.2]
  12 Week Maximum Anal Canal Pressure (Squeeze): number analyzed (Participants) | 68 | 69 | 75 | 37
  12 Week Maximum Anal Canal Pressure (Squeeze) | 83.0 [74.4 to 91.6] | 76.3 [67.7 to 84.9] | 73.6 [65.4 to 81.8] | 73.1 [59.5 to 86.6]
  24 Week Maximum Anal Canal Pressure (Squeeze): number analyzed (Participants) | 70 | 69 | 73 | 35
  24 Week Maximum Anal Canal Pressure (Squeeze) | 83.0 [74.4 to 91.7] | 74.6 [65.9 to 83.4] | 67.1 [58.8 to 75.4] | 72.7 [59.3 to 86.0]

11. Secondary Outcome: Change From Baseline Volume of Air (mL) at First Sensation for Perception of Rectal Distention at 12 and 24 Weeks
Description: Based on data collected from the manometry form, the outcome variable is computed as the difference in volume of air (mL) at first sensation for perception of rectal distention at 12 and 24 weeks and volume of air (mL) at first sensation for perception of rectal distention at baseline.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: volume of air (mL)
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 83 | 81 | 84 | 41
volume of air (mL)
  12 Week Volume of Air at First Sensation: number analyzed (Participants) | 68 | 69 | 76 | 37
  12 Week Volume of Air at First Sensation | 19.0 [14.8 to 23.1] | 22.7 [18.5 to 26.9] | 21.6 [17.6 to 25.5] | 25.1 [18.6 to 31.6]
  24 Week Volume of Air at First Sensation: number analyzed (Participants) | 70 | 69 | 73 | 36
  24 Week Volume of Air at First Sensation | 20.1 [15.9 to 24.3] | 24.5 [20.3 to 28.7] | 21.6 [17.6 to 25.6] | 23.5 [17.1 to 29.8]

12. Secondary Outcome: Change From Baseline Volume of Air (mL) at Urge to Defecate at 12 and 24 Weeks
Description: Based on data collected from the manometry form, the outcome variable is computed as the difference in maximum tolerable rectal volume of air (mL) at 12 and 24 weeks and maximum tolerable rectal volume of air (mL) at baseline.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: volume of air (mL)
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 83 | 81 | 84 | 41
volume of air (mL)
  12 Week Volume of Air at Strong Urge: number analyzed (Participants) | 67 | 68 | 74 | 36
  12 Week Volume of Air at Strong Urge | 69.3 [61.1 to 77.5] | 66.9 [58.7 to 75.2] | 73.0 [65.1 to 80.8] | 71.8 [58.9 to 84.6]
  24 Week Volume of Air at Strong Urge: number analyzed (Participants) | 69 | 68 | 73 | 36
  24 Week Volume of Air at Strong Urge | 76.0 [67.8 to 84.2] | 78.4 [70.0 to 86.7] | 77.3 [69.3 to 85.3] | 73.1 [60.4 to 85.7]

13. Secondary Outcome: Change From Baseline Maximum Anal Pressures During Squeeze With the Catheter at the HPZ at 12 and 24 Weeks
Description: Based on data collected from the manometry form, the outcome variable will be computed as the difference in maximum anal pressures during squeeze with the catheter at the high pressure zone (HPZ) at 12 and 24 weeks and maximum anal pressures during squeeze with the catheter at the HPZ at baseline.
Time Frame: 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: max. anal canal pressure squeeze (mmHg)
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
Number analyzed (Participants) | 83 | 83 | 84 | 41
max. anal canal pressure squeeze (mmHg)
  12 Week Maximum Anal Canal Pressure (Squeeze): number analyzed (Participants) | 68 | 69 | 75 | 37
  12 Week Maximum Anal Canal Pressure (Squeeze) | 83.0 [74.4 to 91.6] | 76.3 [67.7 to 84.9] | 73.6 [65.4 to 81.8] | 73.1 [59.5 to 86.6]
  24 Week Maximum Anal Canal Pressure (Squeeze): number analyzed (Participants) | 70 | 69 | 73 | 35
  24 Week Maximum Anal Canal Pressure (Squeeze) | 83.0 [74.4 to 91.7] | 74.6 [65.9 to 83.4] | 67.1 [58.8 to 75.4] | 72.7 [59.3 to 86.0]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: All events reported by the participants at study visits and EMR review from randomization until 24 weeks
Arm/Group | Loperamide - Exercise Plus Biofeedback | Placebo - Exercise Plus Biofeedback | Loperamide - Education Only | Placebo - Education Only
All-Cause Mortality (participants affected / at risk) | 0/86 | 1/84 | 0/88 | 0/42
Serious Adverse Events (participants affected / at risk) | 6/86 | 5/84 | 10/88 | 3/42
Other Adverse Events (participants affected / at risk) | 71/86 | 60/84 | 60/88 | 26/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loperamide - Exercise Plus Biofeedback (N=86) | Placebo - Exercise Plus Biofeedback (N=84) | Loperamide - Education Only (N=88) | Placebo - Education Only (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loperamide - Exercise Plus Biofeedback (N=86) | Placebo - Exercise Plus Biofeedback (N=84) | Loperamide - Education Only (N=88) | Placebo - Education Only (N=42)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 6 (6) | 6 (7) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5) | 7 (9) | 5 (5)
Constipation (Gastrointestinal disorders) | 44 (61) | 19 (22) | 33 (42) | 5 (8)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (6) | 6 (6) | 7 (8)
Haemorrhoids (Gastrointestinal disorders) | 2 (3) | 5 (5) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (5) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (10) | 10 (11) | 9 (14) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 7 (7) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 2 (3) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No